CLINICAL TRIAL: NCT07337460
Title: Icaritin Soft Capsules Combined With Postoperative Adjuvant Hepatic Arterial Infusion Chemotherapy With mFOLFOX in HCC With High-risk Recurrence Factors: A Single-center, Phase II, Single-arm, Prospective Study
Brief Title: Efficacy and Safety of Icaritin Combined With mFOLFOX in Postoperative HCC With High-risk Recurrence Factors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Dousheng Bai, Clinical Professor, Northern Jiangsu People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025ky300
Record Dates: First submitted 2025-12-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular Carcinoma; postoperative adjuvant chemoinfusion; recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Icaritin Soft Capsules and mFOLFOX-HAIC (Experimental): Treatment:Icaritin Soft Capsules and postoperative adjuvant transarterial chemoinfusion with mFOLFOX
  Interventions: Drug: Icaritin Soft Capsules and mFOLFOX ：Oxaliplatin,leucovorin calcium,5-fluorouracil

INTERVENTIONS:
Drug: Icaritin Soft Capsules and mFOLFOX ：Oxaliplatin,leucovorin calcium,5-fluorouracil — Postoperative adjuvant transarterial chemoinfusion with mFOLFOX.mFOLFOX-HAIC: Oxaliplatin 85 mg/m²via arterial infusion for 2-3 hours, leucovorin calcium 400 mg/m² for 1-2 hours, followed by a 400 mg/m²arterial infusion of 5-fluorouracil for 5 minutes , and continuous arterial infusion at 2400 mg/m²for 46 hours.Within two weeks after the first HAIC procedure, patients should begin taking 2400mg of Icaritin Soft Capsules twice daily for three months, with the total treatment duration not exceeding one year.A second HAIC session was administered 3 weeks later, depending on individual patient conditions, with a maximum of two treatments.

SUMMARY:
This is a single-center, single-arm, prospective trial to explore the efficacy and safety of Icaritin Soft Capsules combined with postoperative adjuvant hepatic arterial infusion chemotherapy(HAIC) with Modified Folinic acid, Fluorouracil, and Oxaliplatin (mFOLFOX) in hepatocellular carcinoma (HCC) with high-risk recurrence factors.

DETAILED DESCRIPTION:
Patients meeting the study's inclusion criteria were enrolled, and their baseline demographic data were collected. Patients enrolled in this study received a first HAIC treatment (mFOLFOX-HAIC) 4-8 weeks after radical surgery. Within two weeks after the first HAIC procedure, patients should begin taking 2400mg of Icaritin Soft Capsules twice daily for three months, with the total treatment duration not exceeding one year. A second HAIC session was administered 3 weeks later, depending on individual patient conditions, with a maximum of two treatments. The protocol specified: Oxaliplatin 85 mg/m²via arterial infusion for 2-3 hours, leucovorin calcium 400 mg/m² for 1-2 hours, followed by a 400 mg/m²arterial infusion of 5-fluorouracil for 5 minutes , and continuous arterial infusion at 2400 mg/m²for 46 hours.

Follow-up was conducted every 8-12 weeks until 12 months postoperatively or the termination of the study. The follow-up included the patient's survival status, tumor recurrence, adverse drug reactions,living quality, routine blood tests, liver function, and electrocardiogram.Contrast-enhanced abdominal CT (layer thickness ≤5 mm) or contrast-enhanced MRI (including DWI sequence) were used for tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤75 years.
2. Histologically/cytologically confirmed hepatocellular carcinoma (HCC) (fibrotic HCC and mixed HCC/biliary carcinoma subtypes were excluded from inclusion criteria), with no prior treatment for HCC (including but not limited to chemotherapy, targeted therapy, immunotherapy, cell therapy, local radiotherapy, and interventional therapy) before surgery.
3. Patients who underwent radical surgery within the first 8 weeks and meet the following criteria: a. Histologically confirmed negative surgical margins (R0) for radical surgery: 1) No residual cancer on gross intraoperative or postoperative imaging; 2) Liver margins>1cm from tumor boundary, or margins ≤1cm with no tumor cell remnants in resected pathological tissue; b. Imaging examination (enhanced chest CT, abdominal CT or MRI, pelvic CT or MRI) performed ≥4 weeks after surgical resection or ablation to confirm complete radiological response.
4. ECOG score ranges from 0 to 1.
5. Patients meeting any of the following high-risk factors for hepatocellular carcinoma recurrence after radical surgery: 1) Single tumor>5 cm 2) Concurrent vascular invasion (microvascular invasion or major vessel invasion Vp1-2) 3) Multiple lesions with ≥3 tumors 4) Tumor grade Edmondson III-IV 5) Surgical margin ≤1cm
6. For patients with preoperative AFP elevation, post-radical surgery or ablation, AFP levels must have significantly decreased and show no significant upward trend.
7. Subjects with Hepatitis B or C Virus(HBV or HCV) infection must undergo standardized antiviral therapy prior to enrollment and continue the treatment during the study period.
8. The patient must have adequate organ and bone marrow function, with laboratory test values meeting the following criteria: 1) Complete blood count (CBC): Absolute neutrophil count (ANC) ≥1.5×10⁹/L; platelet count (PLT) ≥80×10⁹/L; hemoglobin (Hb) ≥90 g/L; 2) Liver function: Serum totalbilirubin (TBIL) ≤2×upper limit of normal (ULN), or direct bilirubin ≤ULN for subjects with TBIL>2×ULN; alanineaminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN; serum albumin ≥28 g/L; 3) Renal function: Serum creatinine (Cr) ≤1.5×ULN, or creatinine clearance (CCr) ≥45 mL/min (Cockcroft-Gault formula) for subjects with Cr>1.5×ULN; 4) Urinalysis shows urine protein <2+; For subjects with baseline urinalysis showing proteinuria ≥2+ in routine urine tests, 24-hour urine collection should be performed with 24-hour urine protein quantification <1g; 5) Coagulation function: International Normalized Ratio (INR) or Activated Partial Thromboplastin Time (APTT) ≤1.5×Upper Limit of Normal (ULN).
9. Life expectancy exceeding 12 months.
10. Not pregnant.

Exclusion Criteria:

1. Presence of extrahepatic metastasis, residual lesions, or recurrence on imaging after surgery or ablation.
2. Patients who have undergone adjuvant therapies such as transarterial chemoembolization (TACE) after radical surgery.
3. Child-Pugh classification grade B or C, or a history of hepatic encephalopathy.
4. Presence of clinically significant pericardial effusion; or clinical symptoms requiring drainage of pleural effusion or ascites.
5. History of bleeding events within 6 months prior to enrollment, such as esophageal or gastric variceal bleeding caused by portal hypertension. Subjects with esophageal or gastric varices requiring intervention within 28 days before enrollment. Untreated or inadequately treated esophageal or gastric varices deemed by investigators to pose a high risk of bleeding.
6. The subject is unable to undergo contrast-enhanced liver CT or MRI scans.
7. Patients who do not meet the criteria for radical surgery.
8. Received Chinese herbal medicine or Chinese patent medicine with antitumor indications or immunomodulatory drugs (including systemic use of thymosin, interferon, etc.) within 14 days prior to enrollment.
9. Participation in other drug clinical trials within 4 weeks prior to enrollment.
10. Co-infection with HBV and HCV (defined as HCV infection history with negative HCV RNA, which was considered as non-infection in this study).
11. History of arterial or venous thromboembolic events occurring within 6 months prior to enrollment, including myocardial infarction (MI), unstable angina, cerebrovascular accident or transient ischemic attack (TIA), pulmonary embolism (PE), deep vein thrombosis (DVT), or any other severe thromboembolic event.
12. Patients with cardiopulmonary insufficiency.
13. Severe infection in the active phase or with poor clinical control. A severe infection within 4 weeks prior to the first treatment, including but not limited to hospitalization due to infection, bacteremia, or severe pneumonia complications.
14. Known hypersensitivity to any investigational drug ingredients; or a history of severe allergic reactions to other traditional Chinese patent medicines.
15. Known history of drug abuse, alcoholism, or substance use.
16. Individuals with a history of psychiatric disorders and lacking capacity for conduct or having limited capacity for conduct.
17. Other acute or chronic diseases, mental disorders, or abnormal laboratory test results that may lead to the following outcomes: increased risks for the subject to participate in the study or receive study treatment, interference with the interpretation of study results, or, at the investigator's discretion, that participation in the study is not in the subject's best interest.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | 2 years
  Recurrence-free survival

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  Overall survival
Time to recurrence (TTR) | 2 years
  Time to recurrence
Safety:treatment-related adverse events (AE) rates | 2 years
  Safety:treatment-related adverse events (AE) rates
living quality | 3 months
  Patient quality of life was evaluated with European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire- Hepatocellular Carcinoma 18(EORTC QLQ-HCC18 )scale.Standardized scores (range: 0-100) were calculated, where increased scores correspond to worse outcomes (i.e., more severe symptoms or impaired quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Dou-sheng Bai, Study Chair — Clinical Medical College, Yangzhou University
Locations (1):
- Clinical Medical College of Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No